CLINICAL TRIAL: NCT02144051
Title: A Phase I, Open-Label, Multicentre Dose-Escalation Study to Investigate the Safety and Pharmacokinetics of AZD5312 in Patients With Advanced Solid Tumours Where the Androgen Receptor Pathway is a Potential Factor
Brief Title: Phase I Open Label Dose Escalation Study to Investigate the Safety & Pharmacokinetics of AZD5312 in Patients With Androgen Receptor Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5860C00001
Record Dates: First submitted 2014-04-29; First posted 2014-05-21 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Advanced Solid Tumours With Androgen Receptor Pathway as a Potential Factor
Keywords: solid tumor, prostate cancer, breast cancer, bladder cancer, ovarian cancer, gastric cancer, salivary duct cancer
MeSH Terms: conditions — Prostatic Neoplasms; Breast Neoplasms; Urinary Bladder Neoplasms; Ovarian Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD5312 (Experimental): AZD5312 will be given intravenously (IV) as an infusion, over one hour. For the purpose of planning, each 4 week period (28 days) will be called a Cycle. AZD5312 will initially be administered 4 times within the first 11 days, (on Days [1, 4, 8 and 11]± 2), with no dosing on sequential days. Patients will receive weekly treatments on Days 15 and 22 to complete Cycle
  1. During the subsequent cycles, patients will receive weekly treatment on Days 1, 8, 15 and 22 (±2).
  Interventions: Drug: AZD5312

INTERVENTIONS:
Drug: AZD5312 — AZD5312 is a generation 2.5 antisense oligonucleotide (ASO) which is designed with the purpose of specifically suppressing human Androgen Receptor (AR) expression, thereby providing potential therapeutic benefit for the treatment of mCRPC and other AR-dependent cancers.
  Other Names: ISIS 560131

SUMMARY:
This is a first time in man (FTIM), Phase I study to determine the Maximum Tolerated Dose, Recommended Phase 2 Dose, safety, tolerability and Pharmacokinetics of AZD5312. This is a multicentre study with sites in the United States and United Kingdom. Approximately 90 patients are expected to be enrolled in this study.

The study involves two parts, Part A, Dose Escalation and Part B, Dose Expansion.

DETAILED DESCRIPTION:
This is a first time in man (FTIM), Phase I study to determine the Maxiimum Tolerated Dose, Recommended Phase 2 Dose, safety, tolerability and Pharmacokinetics of AZD5312. This is a multicentre study with sites in the United States and United Kingdom. Approximately 90 patients are expected to be enrolled in this study.The study involves two parts, Part A, Dose Escalation and Part B, Dose Expansion.

AZD5312 will be given intravenously (IV) as an infusion, over one hour. For the purpose of planning, each 4 week period (28 days) will be called a Cycle. AZD5312 will initially be administered 4 times within the first 11 days, (on Days [1, 4, 8 and 11]± 2), with no dosing on sequential days. Patients will receive weekly treatments on Days 15 and 22 to complete Cycle.

1. During the subsequent cycles, patients will receive weekly treatment on Days 1, 8, 15 and 22 (±2). The AZD5312 dose will not change unless dose reductions are required due to treatment-related toxicity. Patients will continue to receive AZD5312 until disease progression, intolerable toxicity, or discontinuation criteria have been met. Toxicity, Pharmacokinetics and biomarker data will be assessed throughout the study. Alternative infusion durations and/or treatment schedules may be explored if preliminary data suggest these would be more appropriate.

ELIGIBILITY:
Inclusion criteria.

* Patient must understand nature of trial and provide a signed and dated, written informed consent form prior to study specific procedures, sampling and analyses. If a patient declines to participate in voluntary exploratory research and/or genetic component of study, there will be no penalty or loss of benefit to the patient and he/she will not be excluded from other aspects of the study.
* Part A Dose Escalation Patients must have histological or cytological confirmation of a solid tumour of either locally advanced or metastatic castrate resistant prostate cancer (mCRPC), breast, bladder, ovarian, gastric or salivary duct carcinoma where an Androgen Receptor pathway may be a potential factor.
* Part B Dose Expansion.

  * Patient must understand nature of trial and provide a signed and dated, written informed consent form prior to any study specific procedures, sampling and analyses.
  * Part A Dose Escalation Patients must have histological or cytological confirmation of a solid tumour of either locally advanced or metastatic castrate resistant prostate cancer (mCRPC), breast, bladder, ovarian, gastric or salivary duct carcinoma where an Androgen Receptor pathway may be a potential factor.
  * Part B Dose Expansion Arm 1 and 2 patients must have histological or cytological confirmation of locally advanced or metastatic castrate resistant prostate cancer who have progressive disease at the time of entry demonstrated either by Response Evaluation Criteria in Solid Tumors (RECIST) (measurable disease) or by two subsequently increasing Prostate-specific antigen (PSA) values obtained at least one week apart. Arm 3 will include non-mCRPC patients. The patient populations in the dose expansion phase will be as follows:
* Arm 1 Prostate cancer patients with prior second generation anti-hormonal therapy (examples: abiraterone, enzalutamide, TAK 700) without response (disease progression in ≤4 months or Stable Disease (SD) but Prostate-specific antigen (PSA) level did not decline ≥50%).
* Arm 2 Prostate cancer patients with intial response to second generation anti-hormonal therapy (examples: abiraterone, enzalutamide, TAK 700), but later relapsed. Disease relapse would be defined as progressive disease at the time of entry demonstrated either by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 (measurable disease) or by two subsequently increasing Prostate-specific antigen (PSA) values obtained at least one week apart. If clinically meaningful benefits have been identified in a non-mCRPC patient population during the escalation phase, a potential third expansion arm may be considered.
* Arm 3 Patients with a non-mCRPC type solid tumour such as locally advanced or metastatic breast, bladder, ovarian, gastric or salivary duct carcinomas.
* Aged at least 18 years
* Adequate organ system functions, as outined below - Absolute neutrophil count (ANC) ≥1.5 X109/L - Platelets ≥100 X109/L - Haemoglobin ≥9g/dL - aPTT ≤1.5 x ULN - Total bilirubin ≤1.5 mg/dL - Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3.0 times the upper limit of normal (ULN) if no liver involvement or ≤5 times the ULN with liver involvement. - Creatinine ≤1.5 x ULN, OR calculated or measured creatinine clearance ≥50 mL/min as calculated by the Cockcroft-Gault method, OR 24-hour measured urine creatinine clearance ≥50 mL/min.
* Patients must exhibit Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Predicted life expectancy ≥12 weeks
* Patients should have willingness to comply with the study and follow up.
* Male patients with female partners of childbearing potential should be willing to use two forms of acceptable contraception, including one barrier method, during their participation in this study and for 3 months following the last dose of the study drug. Male patients must refrain from donating sperm during their participation in the study and at least for 3 months after the last treatment.
* Female patients should be using adequate contraceptive measures (see Section 3.3). All methods of contraception (with the exception of total abstinence) should be used in combination with the use of a condom by their male sexual partner for intercourse. Female patients should not be breast-feeding and must have a negative pregnancy test prior to start of dosing if of child-bearing potential or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening: - Post-menopausal women defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatment. - Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.

Exclusion criteria

* Patients who have been treated with most recent chemotherapy or investigational drugs ≤21 days or 5 half-lives (whichever is longer) for enrolment, and/or who have National Cancer Institute (NCI) Common Terminology Criteria of Adverse Events (CTCAE) v4.03 Grade 1 treatment-related side effect, with the exceptions of alopecia, should not be enrolled. For further details, please refer to the following link: http://evs.nci.nih.gov/ftp1/CTCAE/About.html.
* Patients who received chemotherapy regimens given either continuously or weekly with limited potential for delayed toxicity or palliative/focal radiotherapy within the last 2 weeks or any other radiotherapy or immunotherapy within 3 weeks of the first dose of study treatment.
* Major surgery (excluding placement of vascular access) ≤21 days of beginning of the study drug or minor surgical procedures ≤7 days. No waiting required following port-a-cath placement.
* Any of the following cardiac criteria: - Congestive heart failure (CHF) per New York Heart Association (NYHA) classification > Class II (see Appendix C) - Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy - Unstable angina or new-onset angina - QTcF >470 ms on screening electrocardiogram (ECG) by Fredericia's formula.
* Patients with leptomeningeal metastases
* Previously untreated brain metastases. Patients who have received radiation or surgery for brain metastases are eligible if therapy was completed at least 3 weeks previously and there is no evidence of central nervous system disease progression, mild neurologic symptoms, and no requirement for chronic corticosteroid therapy.
* As judged by the investigator, any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension, active bleeding diatheses, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required.
* Concurrent conditions that in investigator's opinion would jeopardize compliance with protocol.
* Psychological, familial, sociological, or geographical conditions that do not permit compliance with protocol.

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose of AZD5312 in pts with advanced solid tumours where androgen receptor pathway is a potential factor. | 13 months
  The patient population used for determination of the MTD will consist of patients who have met the minimum safety evaluation requirements of the study, and/or who have experienced a DLT. Minimum safety requirements will be met if, during Cycle 1 of treatment, the patient receives all doses of AZD5312, completes all required safety evaluations, and is observed for at least 28 days following the first dose of AZD5312.
Safety and tolerability of AZD5312 in patients assessed in terms of AEs, labs, vitals, ECGs and conc. med use. | 13 months
Recommended Phase 2 Dose of AZD5312 in patients with advanced solid tumours where androgen receptor pathway is a potential factor. | 13 Months
  •3 evaluable patients (pts) will be enrolled at each dose level (3+3 design) •Evaluated for 28 days before escalation to next dose level. •If more than 1 experiences Dose Limiting Toxicity (DLT), additional 3 patients treated with the same dose. •Maximum of 6 pts enrolled per dose level. •100% increase in dosing until 2 pts (out of 3) at dose level experience toxicity of ≥ Grade 2, or 1 pt. experiences DLT. •Accelerated titration stopped, and subsequent dose escalation will be ≤ 50%. •Evaluation of a cohort of at least 3 patients completing 1 cycle of treatment (28 days) required prior to next dose level. •Dose escalation decisions take into account safety profile of prior dose groups, and available PK data. •Additional patients may be enrolled at lower doses for sufficient PK data. •Intermediate dose levels evaluated to declare the recommended Phase II dose (RP2D). When R2PD is determined, 12 patients will be treated at that dose level to further evaluate safety and efficacy.

SECONDARY OUTCOMES:
Preliminary anti-tumour activity of AZD5312 in patients with advanced solid tumours. | 25 months
  •Proportion of mCRPC patients with a Prostate-specific antigen (PSA) response: Effect of AZD5312 on the PSA levels will be done by looking at PSA by waterfall plots according to the PCWG2 guidelines which measures (1) the percent difference from baseline at 12 weeks treatment points and (2) maximum decline in PSA at any point. •CTC conversions: For prostate cancer patients only, CTC conversions will be asessed which is defined as a significant change in CTC count from the baseline assessment. (Assess absolute reduction in CTC counts). •Metastatic bone disease status of mCRPC patients (PCWG2 criteria, (Scher et al, 2008). •Malignant soft tissue response rate will be assessed byResponse Evaluation Criteria in Solid Tumors (RECIST v1.1) (Eisenhauer et al. 2009) for all patients with measurable disease whenever possible.
Pharmacokinetics of AZD5312 determined by Cmax | 25 months
Pharmacokinetics of AZD5312 determined by tmax | 25 months
Pharmacokinetics of AZD5312 determined by λz | 25 months
Pharmacokinetics of AZD5312 determined by t½λz | 25 months
Pharmacokinetics of AZD5312 determined by (AUC(0-24) | 25 months
Pharmacokinetics of AZD5312 determined by AUC(0-t) | 25 Months
Pharmacokinetics of AZD5312 determined by AUC | 25 months
Pharmacokinetics of AZD5312 determined by CL | 25 months
PK of AZD5312 determined Vz | 25 months
Pharmacokinetics of AZD5312 determined by MRT | 25 Months
Pharmacokinetics of AZD5312 determined by CLR | 25 Months
Pharmacokinetics of AZD5312 determined by Ae;%dose | 25 Months
Pharmacokinetics of AZD5312 determined by Css max | 25 Months
Pharmacokinetics of AZD5312 determined by tss max | 25 Months
Pharmacokinetics of AZD5312 determined by Css min | 25 Months
Pharmacokinetics of AZD5312 determined byAUCss | 25 Months
Pharmacokinetics of AZD5312 determined by CLss | 25 Months
Pharmacokinetics of AZD5312 determined by RAC | 25 Months

CONTACTS AND LOCATIONS:
Overall Officials: Howard Burris, MD, Principal Investigator — SCRI Development Innovations, LLC
Locations (4):
- United States (3):
  - Research Site, Sarasota, Florida
  - Research Site, Nashville, Tennessee
  - Research Site, Milwaukee, Wisconsin
- Research Site, London, United Kingdom